CLINICAL TRIAL: NCT05141591
Title: The Impact of Gender-specific Preoperative Anxiety Level on Postoperative Opioid Requirement After ENT Surgery.
Brief Title: Gender-specific Preoperative Anxiety Level and Postoperative Opioid Requirement After ENT Surgery.
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Other Study IDs: 2006/2021
Record Dates: First submitted 2021-11-10; First posted 2021-12-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Acute Post Operative Pain
Keywords: catastrophizing; opioid consumption
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ENT surgical patients: ASA physical status I-IV adult subjects, ≥ 18 years of age, scheduled for elective ENT surgeries in the Department of ENT at the Medical University of Vienna. On the day before elective ENT- surgery patients will be asked to complete self-administered questionnaires (STOA, APAIS, PCS) concerning their emotional and anxiety state. These questionnaires will be re-tested on the day of surgery and opioid consumption during the stay in the recovery room documented.
  Interventions: Other: Anxiety level assessment

INTERVENTIONS:
Other: Anxiety level assessment — To investigate the impact of psychological variables e.g. pre-surgical anxiety on postoperative opioid consumption and pain level, the investigators will perform the STOA, APAIS, PCS and the VAS-A anxiety questionnaires before surgery.

SUMMARY:
The study will be designed to investigate the impact of the preoperative anxiety level on postoperative opioid requirement during the PACU stay, in order to improve postoperative pain treatment in the long term after ENT surgery.

The present study can contribute to improve postoperative pain management in patients in the field of ENT surgery, as new influencing parameters and risk factors may be discovered.

DETAILED DESCRIPTION:
Background Due to the frequency of surgeries, acute postsurgical pain (APSP) is a common clinical problem. In this study, the investigators will investigate pre-surgical psychological factors associated with the experience of APSP in ENT surgery.

The study will be designed to investigate the impact of gender-specific preoperative anxiety states, using the STOA, APAIS, PCS and VAS-A scoring systems, on postoperative opioid consumption after elective ENT surgery.

These findings may have important implications for developing more personalized strategies in acute postoperative pain therapy in selected patients.

Aim Study aim is to investigate the impact of the preoperative anxiety level, using the validated STOA questionnaire, on postoperative opioid requirement during the PACU stay, in order to improve postoperative pain treatment in the long term after ENT surgery.

The present study can contribute to improve postoperative pain management in patients in the field of ENT surgery, as new influencing parameters and risk factors may be discovered.

The investigators hypothesize that a higher preoperative anxiety state, is a predictive factor of opioid requirement in the early postoperative period after ENT surgery.

Methods Surgery-related psychological factors like anxiety state will be assessed gender-specific, in patients scheduled for elective ENT surgery by validated questionnaires (STOA, APAIS, PCS and VAS-A), filled out by the patient the day before surgery and on the day of surgery, to investigate the correlation with the postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-IV
* able to read and understand the information sheet and to sign the consent form
* being scheduled for elective ENT surgery under general anesthesia
* written informed consent
* age≥18 years

Exclusion Criteria:

* difficulty to understand study procedure, pain scoring system or questionnaires
* surgical procedure warranting elective postoperative ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will study ASA physical status I-IV adult subjects, ≥ 18 years of age, scheduled for elective ENT surgeries in the Department of ENT at the Medical University of Vienna. Written informed consent will be obtained from each participant.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | during the stay in the recovery room assessed up to 2 hours
  cumulative opioid consumption within PACU stay

SECONDARY OUTCOMES:
Postoperative Pain Score-VAS-PACU | during the stay in the recovery room assessed up to 2 hours
  mean pain level on an 11-point verbal Likert response score recorded at 30-minute intervals during the PACU stay, ranging between 0 and 10, with higher levels indicating higher pain intensity

OTHER OUTCOMES:
Anxiety scores-APAIS | on the 1 day before surgery and on the 1 day of surgery
  APAIS-Amsterdam Preoperative Anxiety and Information Scale Total range 6 to 30, a higher value reflects a higher anxiety as well as higher information requirement.
Postoperative Pain Score-VAS | during the stay in the recovery room assessed up to 2 hours
  NRS score: evaluated at arrival and discharge from the PACU time to first analgesic (non-opioid, opioid) supplementation postoperatively in the PACU
Anxiety scores-PCS | on the 1 day before surgery and on the 1 day of surgery
  PCS-Pain catastrophizing scale The higher the total score, the greater the individual risk of catastrophic pain. The PCS score ranges from 0 to 52 points.
VAS-A. anxiety score | preoperative on the 1 day of surgery, immediately postoperative in the PACU
  The VAS-A scale is comprised of a horizontal line 100mm long with the indication "no anxiety" to the left and "worst possible anxiety" to the right. The higher the total score, the greater the individual anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria